CLINICAL TRIAL: NCT01138059
Title: REperfusion Therapy in Acute Ischemic STroke With Unclear Onset by MRI Evaluation
Brief Title: Reperfusion Therapy in Acute Ischemic Stroke With Unclear Onset
Acronym: RESTORE
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Dong-Wha Kang, Asan Medical Center
Other Study IDs: AMC-2004-217
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2006-10

CONDITIONS: Stroke
Keywords: Acute ischemic stroke with unclear onset time
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute ischemic stroke patients with unclear onset

SUMMARY:
This study will test the hypothesis whether patients with unclear-onset stroke (UnCLOS) treated with thrombolysis could achieve a prespecified rate of good clinical outcome. The secondary hypothesis is that the efficacy outcomes in UnCLOS group would be superior to those in historical UnCLOS group from prospective stroke registries.

DETAILED DESCRIPTION:
1. Study design: A prospective multicenter trial
2. Study centers: 6 participating medical centers in South Korea
3. Participants: Consecutive patients with acute ischemic stroke visiting the emergency room within 6 hours of the detection of stroke symptoms
4. Methods

   * 3 thrombolysis protocols applicable to UnCLOS patients

     1. IV tissue plasminogen activator (tPA) : Conventional intravenous tPA (0.9 mg/kg, 10% of the dose as a bolus and the remainder over 60 minutes) will be administered to patients within 3 hours of first found abnormal time who had no arterial occlusion or catheter-inaccessible occlusion.
     2. IV tPA + IA urokinase protocol : Combined intravenous tPA (0.6 mg/kg, 10% of the dose as a bolus and the remainder over 30 minutes) with intra-arterial urokinase will be administered to those within 3 hours from first found abnormal time who had catheter-accessible arterial occlusion.
     3. IA UK protocol : Intra-arterial urokinase will be given to those between 3 and 6 hours after first found abnormal time who had catheter-accessible arterial occlusion.
5. Outcome variables

   * Safety outcomes Symptomatic intracranial hemorrhage (ICH) within 48 hours from thrombolytic therapy.
   * Efficacy outcomes

     1. Long-term clinical outcomes (modified Rankin Scale) at 3 months
     2. Secondary efficacy outcomes : Good vs. Poor outcomes according to mRS responder analysis, Early neurological improvement, Immediate and 5-day recanalization on MRA or CTA

ELIGIBILITY:
Inclusion Criteria:

1. The patient is male or female and age between 18 and 85 years
2. The patient has unclear onset stroke
3. Treatment of the patient can be initiated within 6 hours after first found abnormal time
4. The patient has imaging-defined penumbra (at least 20%), measured by diffusion- and perfusion-weighted MRI

Exclusion Criteria:

1. The patient has minor neurologic deficits (NIHSS <4, except aphasia or hemianopia).
2. The patient has rapidly resolving neurological symptoms and the rate of improvement is projected to give the patient an NIHSS score <4 at the time of treatment.
3. The patient has a pre-stroke mRS score of >1 (indicating previous disability).
4. The symptoms of stroke are suggestive of subarachnoid hemorrhage.
5. Evidence of infective endocarditis or septic embolism
6. The patient has a history or clinical presentation of ICH, SAH, or AVM.
7. Serious head trauma within 6 weeks
8. Prior ischemic stroke in previous 6 weeks (except small infarct)
9. Myocardial infarction in the previous 3 weeks
10. Gastrointestinal or urinary tract bleeding in previous 21 days
11. Major surgery in the previous 14 days
12. History of biopsy of a parenchymal organ, trauma with internal organ injury or lumbar puncture within 14 days
13. Arterial puncture at a non-compressible site in the previous 7 days
14. Uncontrolled high blood pressure (systolic > 185 mmHg or diastolic > 110 mmHg on 3 separate occasions at least 10 min apart despite appropriate treatment)
15. Evidence of active bleeding or acute trauma (fracture) on examination
16. Current use of oral anticoagulants and a prolonged prothrombin time (INR >1.7)
17. The patient has been treated with heparin in the previous 48 hours with prolonged aPTT, except for low dose subcutaneous LMWH with doses recommended for DVT prophylaxis
18. Baseline platelet count < 100,000 mm3
19. Baseline hematocrit < 25%
20. Blood glucose concentration < 50 mg/dL (2.7 mmol/L) in case of CT screening
21. Seizure at onset with postictal residual neurological impairments in case of CT screening
22. The patient has a terminal illness.
23. The patient is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.
24. The patient has extensive early infarction in any affected area defined as an infarcted core involving > 1/3 of MCA territory or the entire ACA or PCA territory
25. The patient has well-developed parenchymal hyperintensity on FLAIR, T2*, or EPI-T2 images, or marked hypodensity on CT, indicative of subacute infarction, or enhancement with morphologic features suggesting the lesion is more than 6 hours old
26. The patient has a contraindication to the imaging techniques (this means ferromagnetic objects for MRI, contraindications to contrast agent, renal disease with iodinated contrast agent in perfusion CT and CTA, etc.)
27. The patient has imaging evidence of ICH or SAH, AVM, brain tumor (Incidental meningioma and microbleeds are not exclusion criteria. Incidental unruptured aneurysm that is small (< 5mm) is not an exclusion criterion).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute ischemic stroke visiting the ER within 6 hours of the detection of stroke symptoms will be screened for this study.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Good clinical outcome defined as modified Rankin Scale 0-2 | 3 months after treatment
Symptomatic intracranial hemorrhage | 48 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wha Kang, MD, PhD, Principal Investigator — Asan Medical Center